CLINICAL TRIAL: NCT02439034
Title: Paracetamol With or Without Ketoprofen in the Management of Pain During Hospitalisation and at Home for Patients Receiving Brachytherapy: Phase-2 Randomized Study
Brief Title: Paracetamol With or Without Ketoprofen in the Management of Pain for Patients Receiving Brachytherapy (KETOCOL-1304)
Acronym: KETOCOL-1304
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Oscar Lambret (Other)
Collaborators: Santelys Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KETOCOL-1304
Record Dates: First submitted 2015-04-30; First posted 2015-05-08 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-07

CONDITIONS: Uterine Cervical Cancer; Upper Aerodigestive Tract Neoplasms
Keywords: pain management; brachytherapy
MeSH Terms: conditions — Uterine Cervical Neoplasms; Head and Neck Neoplasms; Agnosia | interventions — Acetaminophen; Ketoprofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Active Comparator): Paracetamol
  Interventions: Drug: Paracetamol
- Arm B (Experimental): Paracetamol + Ketoprofen
  Interventions: Drug: Paracetamol; Drug: Ketoprofen

INTERVENTIONS:
Drug: Paracetamol — Paracetamol 1 g IV then 1 g 3 times a day IV or oral (PO)
  Other Names: PARACETAMOL B BRAUN; PARACETAMOL CODEINE ARROW
Drug: Ketoprofen — Ketoprofen* 100 mg (IV then PO) : Ketoprofen 100 mg IV 2 times a day or Ketoprofen LP 100 mg PO 2 times a day.
  Other Names: BI PROFENID LP; PROFENID
  Arms: Arm B

SUMMARY:
The results of the study will permit to set up a standardized and validated procedure of pain management authorizing medical and paramedical staff of brachytherapy department to handle pain and in this way to improve the quality of life of the patients.

DETAILED DESCRIPTION:
* Selection criteria validation
* Patient information and collection of a signed informed consent
* Randomization
* Completion of HADS questionnaire
* Day 1 = Begin of analgesic treatment / brachytherapy
* T-30= 30 minutes before the operative procedure, IV administration of the analgesic treatment (Arm A or B) by the anesthetist
* T0= end of the operative procedure under general anesthesia
* T4, T8, and T12 = 4, 8 and 12 hours after T0: evaluation of pain level. If pain level ≥ 4:

  1. paracetamol-codeine (Arms A and B) and continuation of ketoprofen (Arm B). Then, if persistence of pain :
  2. paracetamol and morphine (Arms A and B)
* Day 2 to Day 30: At home or during hospital stay:

Pain assessment twice a day by the patient until absence of pain during 2 consecutive days

* Day 3 and Day 15: Pain assessment or phone interview by the algologist of the investigation center ; completion of a HADS questionnaire on Day 3
* Day 30= End of study: Pain assessment by the algologist of the investigation center and HADS questionnaire

In any case, pain assessment must be done until absence of pain during 2 consecutive days

ELIGIBILITY:
Inclusion Criteria:

* Patient with a uterine cervical cancer or an upper aero-digestive tract cancer
* Age ≥ 18 years and ≤ 75 years
* Patient who are eligible for brachytherapy treatment associated with or without hospital stay
* With operative procedure under general anesthesia to set up the material needed for brachytherapy
* Performance status ≤ 2
* Creatinine Clearance ≥ 60 ml/min using Cockcroft equation
* No coagulation disorder or anticoagulation therapy at curative dose
* Registered with a social security system
* Patient having dated and signed an informed consent form before initiation of any study procedures

Exclusion Criteria:

* Respiratory pathology (SpO2< 70 %)
* Severe undernutrition
* Previous hypersensitivity reactions such as bronchospasm, asthma, rhinitis, hives or other allergic reaction to ketoprofen, to acetylsalicylic acid, or other NSAIDs
* Previous hemorrhage or gastrointestinal perforation during a previous treatment with NSAID
* Gastrointestinal hemorrhage , cerebrovascular hemorrhage or other evolutive hemorrhage
* Evolutive peptic ulcer, previous peptic ulcer or recurring hemorrhage (2 or more distinct episodes of hemorrhage or ulcer objectified)
* Liver insufficiency
* Severe renal insufficiency
* Severe heart failure
* Treatment with another NSAID, including selective cyclooxygenase-2 inhibitors
* Intolerance or hypersensitivity to one of the treatments or excipients
* Inability to swallow
* Pregnant or breastfeeding woman
* Patient under tutorship or guardianship

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-02; Primary Completion 2018-02 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Level of immediate post-operative pain | Day 1
  Immediate post-operative pain will be assessed on a scale from 0 to 10. Experimental treatment will be considered as a success if the level of pain is < 4, 4 hours after the surgical operation.

SECONDARY OUTCOMES:
Level of pain linked to the operative procedure during brachytherapy and at home | Day 1 (8, 12 hours), Days 3, 15 and 30
  Assessment of the pain level at 8, 12 hours after the operative procedure, then twice a day during hospital stay or at home until the absence of pain during 2 consecutive days. This level will also be measured at days 3, 15 and 30 at hospital or during a phone interview (Days 3 and 15) and by the algologist of the investigation center on Day 30.
Tolerance of the analgesic treatment | 30 days
  assessment based on NCI-CTCAE v4.0
Assessment of anxiety before, during and after brachytherapy by completing the HADS questionnaire | inclusion, Days 3 and 30

CONTACTS AND LOCATIONS:
Overall Officials: Danièle LEFEBVRE-KUNTZ, MD, Study Director — Centre Oscar Lambret; Nathalie LEROUX, MD, Study Director — Centre Oscar Lambret
Locations (1):
- Centre Oscar Lambret, Lille, France

IPD SHARING:
Plan to Share IPD: No